CLINICAL TRIAL: NCT06180057
Title: Randomized, Two-way, Two-period, Single Oral Dose, Open-label, Crossover, Bioequivalence Study to Compare Chenodeoxycholic Acid Capsules (250mg Chenodeoxycholic Acid) [Dose: 1 x 02 Capsules] Versus Chenodeoxycholic Acid Leadiant 250 mg Hard Capsules (250mg Chenodeoxycholic Acid) [Dose: 1 x 02 Capsules] in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study to Compare Chenodeoxycholic Acid Capsules (250mg Chenodeoxycholic Acid) Versus Chenodeoxycholic Acid Leadiant 250 mg Hard Capsules (250mg Chenodeoxycholic Acid)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1164-2022
Record Dates: First submitted 2023-12-05; First posted 2023-12-22 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Cerebrotendinous Xanthomatoses
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous | interventions — Chenodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chenodeoxycholic acid capsules (Experimental): Chenodeoxycholic acid capsules (250mg chenodeoxycholic acid)
  Interventions: Drug: Chenodeoxycholic acid
- Chenodeoxycholic acid leadiant hard capsules (Active Comparator): Chenodeoxycholic acid leadiant hard capsules (250mg chenodeoxycholic acid)
  Interventions: Drug: Chenodeoxycholic acid leadiant

INTERVENTIONS:
Drug: Chenodeoxycholic acid — Two capsules were administered orally
  Arms: Chenodeoxycholic acid capsules
Drug: Chenodeoxycholic acid leadiant — Two capsules were administered orally
  Arms: Chenodeoxycholic acid leadiant hard capsules

SUMMARY:
Randomized, two-way, two-period, single oral dose, open-label, crossover, bioequivalence study to compare Chenodeoxycholic acid capsules (250mg chenodeoxycholic acid) [dose: 1 x 02 capsules] versus Chenodeoxycholic acid leadiant 250 mg hard capsules (250mg chenodeoxycholic acid) [dose: 1 x 02 capsules] in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria

* The subject is Caucasian & aged between eighteen to fifty years (18 - 50), both inclusive.
* The subject is within the limits for his height & weight as defined by the body mass index range (18.5 - 25.0 Kg/m2).
* The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
* The results of medical history, vital signs, physical examination & conducted medical laboratory tests are normal as determined by the clinical investigator.
* The subject tested negative for Hepatitis B (HBsAg), Hepatitis C (HCVAb) and human immunodeficiency virus (HIVAb).
* There is no evidence of psychiatric disorder, antagonistic personality and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* The subject is able to understand and willing to sign the informed consent form.
* For female subjects: negative serum pregnancy test and the woman is using a reliable contraception method.
* The subject has normal cardiovascular system & ECG recording.
* The subject kidney and liver (aminotransferase & Alanine transaminase enzymes) functions tests are within normal range. (Creatinine is accepted if below the reference range after being evaluated by the CI as clinically not significant).
* The subject has normal Triglyceride (0.1-150 mg/dl), HDL (35-55 mg/dl), LDL (0.1-159 mg/dl) and Total Cholesterol levels (0.1-200 mg/dl) or clinical insignificant based on CI evaluation.

Exclusion Criteria

* The subject is a heavy smoker (more than 10 cigarettes per day).
* The subject has suffered an acute illness one week before dosing.
* The subject has a history of or concurrent abuse of alcohol.
* The subject has a history of or concurrent abuse of illicit drugs.
* The subject has a history of hypersensitivity and/or contraindications to the study drug; including its excipients and any related compounds.
* The subject has been hospitalized within three months before the study or during the study.
* The subject is on special diet (for example subject is vegetarian.)
* The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 72 hours after dosing in both study periods.
* The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.
* The subject has taken grapefruit/orange containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.
* The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.
* The subject has donated blood within 80 days before first dosing.
* The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.
* Subject has consumed medicines or foodstuff that may affect pharmacological or pharmacokinetic properties of chenodeoxycholic acid (for example: Antacids (aluminum containing), Bile acid sequestrants such as (cholestyramine or colestipol), Clofibrate, Coumarin-derivative anticoagulants, Estrogens & oral contraceptive) two weeks before dosing, during the study and two weeks after dosing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 72 hours
  Statistical analysis of primary endpoints will include descriptive statistics, Analysis of Variance (ANOVA), and Confidence Interval (CI). The average bioequivalence of the products is concluded if the two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data for Cmax
Area under the plasma concentration-time curve from time 0 to 12 hours (AUC0-12) | 12 hours
  Statistical analysis of primary endpoints will include descriptive statistics, Analysis of Variance (ANOVA), and Confidence Interval (CI). The average bioequivalence of the products is concluded if the two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data for AUC0-12

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to 72 hours (AUC0-72) | 72 hours
  The descriptive statistics for AUC0-72

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- ACDIMA Biocenter, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No